CLINICAL TRIAL: NCT00406835
Title: Phase 3 Study of Whole Brain Radiation Therapy Plus Stereotactic Radiosurgery Versus Stereotactic Radiosurgery Alone for 1-4 Brain Metastases
Brief Title: Prospective Randomized Trial Between WBRT Plus SRS Versus SRS Alone for 1-4 Brain Metastases
Status: Completed | Type: Observational
Sponsor: Hokkaido University Hospital (Other)
Other Study IDs: JROSG99-1
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Brain Metastasis
Keywords: Whole Brain Radiation Therapy; Stereotactic Radiosurgery; Brain metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Whole-Brain Radiation Therapy, Stereotactic Radiosurgery

SUMMARY:
The purpose of this study is to determine if WBRT combined with SRS resulted in improvements in survival, brain tumor control, functional preservation rate, and frequency of neurologic death.

DETAILED DESCRIPTION:
Whole-Brain Radiation Therapy (WBRT) had been a mainstay in the treatment of brain metastases. However, treatment strategy which rely on Stereotactic Radiosurgery (SRS) has becoming popular in Japan. It is not well understood if the Whole-Brain Radiation Therapy (WBRT) combined with Stereotactic Radiosurgery (SRS) resulted in improvements in survival, brain tumor control, functional preservation rate, and frequency of neurologic death. In orer to determine the role of WBRT, we conducted prospective randomized trial between WBRT+SRS and SRS-alone for 1-4 brain metastatic patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with 1-4 brain metastases, each with a maximum diameter of no more than 3 cm on contrast-enhanced MRI scans, and were derived from a histologically confirmed systemic cancer, Karnofsky Performance Status (KPS) score of 70 or more

Exclusion Criteria:

* Patients with metastases from small cell carcinoma, lymphoma, germinoma, and multiple myeloma were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 1999-10; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Hidefumi Aoyama, MD, PhD, Principal Investigator — Hokkaido University School of Medicine; Hiroki Shirato, MD, PhD, Study Chair — Hokkaido University School of Medicine; Keiichi Nakagawa, MD, PhD, Study Director — Tokyo University
Locations (1):
- Hokkaido University School of Medicine, Sapporo, Hokkaido, Japan